CLINICAL TRIAL: NCT06460298
Title: Phase I/II Trial Evaluating the Safety and Efficacy of ProAgio, an Anti- αvβ3 Integrin Cytotoxin, in Combination With Gemcitabine in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: ProAgio in Combination With Gemcitabine in Patients With Metastatic Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ProDa BioTech, LLC (Industry)
Collaborators: Emory University (Other); Georgia State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BIO 01192022
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: This study includes a dose escalation arm, followed by an expansion arm at the ideal dose for participants To estimate the objective response rate (ORR) of ProAgio in combination with gemcitabine in patients with metastatic TNBC who have been previously treated with at least two prior lines of therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Experimental: Dose Escalation ProAgio Dose Levels (DL) 1,2,3,4 ProAgio combined with Gemcitabine is administered to study participants by intravenous injections on days 1, 8, 15, every 4-week Cycle.
  Other Names:
  ACT50, and Gemcitabine
  Interventions: Drug: ProAgio Dose Levels (DL) 1,2,3,4
- Dose Expansion (Experimental): Participants will receive ProAgio at the objective response rate (ORR) combined with Gemcitabine is administered to study participants by intravenous injections on days 1, 8, 15 every 4-week Cycle.
  Other Names:
  ACT50, and Gemcitabine
  Interventions: Drug: ProAgio Dose Expansion

INTERVENTIONS:
Drug: ProAgio Dose Levels (DL) 1,2,3,4 — ProAgio combined with Gemcitabine in patients with metastatic TNBC who have been previously treated with at least two prior lines of therapy.
  Other Names: ACT50; Gemcitabine
  Arms: Dose Escalation
Drug: ProAgio Dose Expansion — ProAgio combined with Gemcitabine in patients with metastatic TNBC who have been previously treated with at least two prior lines of therapy.
  Other Names: ACT50; Gemcitabine
  Arms: Dose Expansion

SUMMARY:
This is a Phase I/II Trial Evaluating the Safety and Efficacy of ProAgio, an anti- αvβ3 Integrin Cytotoxin, in Combination with Gemcitabine in Patients with Metastatic Triple Negative Breast Cancer

DETAILED DESCRIPTION:
This is a single-arm, Phase I/II study, designed to evaluate the safety and efficacy of the combination of ProAgio with gemcitabine in patients with previously treated, metastatic triple negative breast cancer.

Dose escalation will proceed using the Bayesian Optimal Interval (BOIN) design, with a target toxicity rate of 0.25, a maximum sample size of 20, and a cohort size of 2.

There are four dose levels considered in the dose escalation phase, and we start at the lowest dose level (Dose Level 1).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, ≥ 18 years of age, with histologically or cytologically confirmed metastatic breast cancer that is estrogen receptor (ER) negative (less than 10%), progesterone receptor (PR) negative (less than 10%), and HER2 negative/unamplified as per ASCO/CAP guidelines (Wolff et al., 2018). If ER/PR less than 10%, prior endocrine therapy is permitted, and the participant is not considered appropriate for hormone based therapy. Participants must agree to provide archival tumor material from metastatic site (most recent archival tumor tissue immediately prior to enrollment is strongly preferred) and must agree to undergo research tumor biopsy before treatment and during cycle 2 at the same site of metastatic disease, if presence of easily accessible lesion, at the discretion of the treating physician.
* Participants must have received at least two lines of prior systemic treatment for advanced disease. If participants received systemic therapy in the operable setting and the tumor progressed within 12 months of the receipt of the last dose of systemic therapy, this will be considered one line of prior systemic therapy for advance disease. Participants must be more than 14 days removed from most recent standard of care or experimental drug treatment for their tumor.
* ECOG performance status ≤2
* Participants must have adequate organ and marrow function as defined below:
* Absolute neutrophil count ≥1,500/mcL
* Hemoglobin ≥9 g/ dL (recent transfusion allowed)
* Platelets ≥100,000/mcL
* AST(SGOT)/ALT(SGPT) ≤3 x ULN. AST and ALT (up to 5x ULN is permitted for participants with liver metastases)
* Total bilirubin ≤1.5 x institutional ULN
* Creatinine clearance ≥60 mL/min (measured using Cockcroft- Gault equation or the estimated glomerular filtration rate)
* Participants with CNS metastases must be treated and/or stable (no progression for at least 4 weeks after local prior therapy as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period). Those with symptoms suggestive of possible CNS metastases (such as new headaches) must undergo brain MRI as part of screening.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of ProAgio on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for the 6 months following the last dosing of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* During dose escalation, participants with bone only and/or non-measurable disease are eligible. During dose expansion, only participants with measurable disease are eligible.
* Ability of subject to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had prior treatment with gemcitabine in the metastatic setting.
* Platelet transfusion within 7 days prior to treatment start.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better. Patients with history of known congestive heart failure (left ventricular ejection fraction (LVEF) <50%) must have documented LVEF >50% within 12 months of study enrollment.
* Prolonged QTc interval >480 msec on screening EKG
* Participants with known diagnosis of a chronic neurologic disorders (such as multiple sclerosis, Huntington's disease, Parkinson's disease, or uncontrolled epilepsy) which causes motor disturbance, visual disturbance, or seizure and could confound assessment of neurologic toxicity caused by the study drug.
* Pregnant or nursing women are excluded from this study because ProAgio is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ProAgio, breastfeeding should be discontinued if the mother is treated with ProAgio.
* Participants who have undergone a major surgical procedure (within < 28 days) are excluded.
* Participants with uncontrolled bleeding episodes <28 days prior to enrollment are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Dose Escalation) | 2 Years
  To identify the maximum tolerated dose (MTD) of ProAgio in combination with gemcitabine in patients with metastatic TNBC who have been previously treated with at least two prior lines of therapy.
Part 2 (Dose Expansion) | 2 Years
  To estimate the objective response rate (ORR) of ProAgio in combination with gemcitabine in patients with metastatic TNBC who have been previously treated with at least two prior lines of therapy.

SECONDARY OUTCOMES:
Clinical Benefit Rate | 2 Years
  To describe the clinical benefit rate (CBR) in patients with metastatic TNBC treated with ProAgio in combination with gemcitabine.
Estimate the mean change from baseline in tumor stromal collagen | 2 Years
  To estimate the mean change from baseline in tumor stromal collagen following treatment with ProAgio and gemcitabine.
Progression free survival (PFS) | 2 Years
  To describe the progression free survival (PFS) in patients with metastatic TNBC treated with ProAgio in combination with gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kalinsky, M.D, M.S, Principal Investigator — Emory University Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No